CLINICAL TRIAL: NCT01985503
Title: Brown Adipose Tissue: Longitudinal Follow-up of Brown Adipose Tissue Structure and Associations With Obesity and Cardiovascular Risk Factors in Healthy Participants of Baseline PET Studies (BAT-Follow-Up)
Brief Title: Longitudinal Follow-up of Brown Adipose Tissue Function and Structure
Acronym: BATFollowUp
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Juho Raiko, MD, PhD, Turku University Hospital
Other Study IDs: BAT-Follow-Up; BATFOLLOWUP (Other: PET Centre, Turku University)
Record Dates: First submitted 2013-11-04; First posted 2013-11-15 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Obesity
Keywords: positron emission tomography; magnetic resonance imaging; brown adipose tissue; obesity; cardiovascular disease; subclinical atherosclerosis
MeSH Terms: conditions — Obesity; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood samples, fecal samples, adipose tissue biopsies and skeletal muscle biopsies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Phase 1 group: Subjects were studied in 2009 and their follow-up is in 2014.
- Phase 2 group: Subjects were studied in 2011 and their follow-up is in 2016.

SUMMARY:
In Turku PET Centre, there have been 3 positron emission tomography studies on brown adipose tissue (BAT) activity in healthy adults. BATPET was performed between 2008 and 2009. FATBAT started in 2011 and Dixon-BAT in 2012 and they are both currently ongoing. In the current study, participants of BATPET, FATBAT and Dixon-BAT studies are recruited for a follow-up study to examine associations between obesity, cardiovascular risk factors, serum metabolic profile and BAT structure at baseline and during follow-up several years later. 43 BATPET participants will be called for follow-up in 2013 with a follow-up period of 5 years and 52 FATBAT and Dixon-BAT participants in years 2014 and 2015 with a follow-up period of 3 years. The aim of this study is to examine longitudinal associations between BAT function and structure, liver adiposity and cardiovascular risk factors at baseline and during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All study subjects have been screened prior to acceptance in BATPET, FATBAT and Dixon-BAT studies and no screening for inclusion is required in the current study.

Exclusion Criteria:

* 1) Smoking 2) Blood pressure > 160/100 mmHg 3) Pregnancy or lactation 4) Medication (expected effect on study variables)

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study subjects are healthy 22-55-year-old Caucasians. Population contains both lean and obese subjects.
Sampling Method: Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation between baseline brown adipose tissue activity according to PET imaging and serum lipoprotein concentrations at follow-up 5 years later | 5 years
  Brown adipose tissue activity is determined with FDG-PET imaging at baseline in 43 subjects and 5 years later the subjects participate a follow-up visit where lipoprotein levels are measured in mmol/l from serum samples. Correlation between brown adipose tissue activity and serum lipoproteins are examined with Pearson's correlation.

SECONDARY OUTCOMES:
Association between brown adipose tissue structure at baseline and at follow-up | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Juho RH Raiko, MD, PhD, Principal Investigator — PET Centre, Turku Univesity
Locations (1):
- PET Centre, Turku University, Turku, Finland